CLINICAL TRIAL: NCT06746337
Title: IMAGINE: Pilot Trial of a Digital Group Intervention to Prevent Perinatal Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Northwestern University (Other); Brown University (Other); Seattle Children's Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Keshet Ronen, Assistant Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00019195; R34MH131571 (NIH)
Record Dates: First submitted 2024-12-12; First posted 2024-12-24 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Depression During Pregnancy; Depression, Postpartum
Keywords: digital; perinatal; depression
MeSH Terms: conditions — Depression, Postpartum; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMAGINE (Experimental): The intervention is a digital adaptation of the evidence-based Mothers and Babies program, delivered interactively to groups of perinatal people and facilitated by a mental health provider.
  Interventions: Behavioral: IMAGINE
- Control (No Intervention): Control participants will be provided with standardized information about signs and symptoms of perinatal depression and will continue to receive standard healthcare.

INTERVENTIONS:
Behavioral: IMAGINE — IMAGINE is a digital group cognitive behavioral therapy intervention
  Arms: IMAGINE

SUMMARY:
The goal of this clinical trial is to evaluate if a digital group intervention (named IMAGINE) can prevent depression in perinatal populations. The main questions it aims to answer are:

Does IMAGINE engage cognitive behavioral therapy targets? Does IMAGINE lead to lower depression scores? Is IMAGINE acceptable, appropriate, usable and feasible?

Participants will be randomized to either participate in an IMAGINE group for 12 weeks or receive standard of care. Participants will respond to questionnaires at enrollment and study visits at 12 and 24 weeks after enrollment.

DETAILED DESCRIPTION:
Perinatal depression affects an estimated 13% of pregnant people in the US. While effective interventions exist to prevent perinatal depression, access to facility-based in-person interventions is limited. This proposal will refine a digital group adaptation of an evidence-based prevention intervention, and evaluate its preliminary effectiveness and implementation outcomes through a pilot randomized controlled trial.

The proposal consists of 3 specific aims:

Aim 1. Using human-centered design, refine the IMAGINE intervention for implementation within perinatal mental health services in Washington State. Building off existing IMAGINE intervention materials, we will conduct qualitative interviews and focus groups with perinatal people, service providers, administrators, and payers to refine:

1. IMAGINE intervention design to meet the needs of perinatal clients age 16-35. Components to be optimized include message frequency, balance of synchronous and asynchronous content, and group composition.
2. IMAGINE implementation protocols and materials to support delivery by our implementation partner.

Hypothesis: Combined synchronous and asynchronous content and delivery compliant with billable health services will be preferred.

Aim 2. Determine IMAGINE's preliminary effectiveness engaging CBT targets and preventing depression.

A pilot RCT will be conducted comparing IMAGINE (as optimized in Aim 1) delivered in English or Spanish vs. treatment as usual, among 100 perinatal participants (pregnant or ≤6 months postpartum) with one or more risk factors for perinatal depression (as defined by USPSTF) and no current major depression. Participants will be recruited from our partner organization's clients. We will compare longitudinal change in depression symptoms and engagement of target mechanisms (negative mood regulation, perceived stress, and perceived social support) between arms at enrollment, 12- and 24-weeks post-enrollment. Exploratory analyses will assess effect modification by participant age, race/ethnicity, pregnancy status, and language.

Hypothesis: IMAGINE will lead to moderate reduction in depression symptoms, with effect size similar to MB.

Aim 3. Determine IMAGINE's preliminary implementation outcomes (acceptability, appropriateness, usability, and feasibility) among client, provider, administrator, and payer stakeholders.

Acceptability, appropriateness and usability among RCT participants will be assessed based on quantitative questionnaires, engagement in IMAGINE, and qualitative interviews. Provider, administrator, and payer acceptability, feasibility, and appropriateness will be determined through group discussion of IMAGINE RCT process indicators. We will explore client and contextual determinants of implementation outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or up to 6 months postpartum
* Age 16 or over
* At elevated risk of perinatal depression (per USPSTF)
* Speaks English or Spanish
* PHQ9<15 and no current major depression
* Access to a smartphone with cellular data at least 3 days per week
* If receiving other mental healthcare services, has been established in care at least 6 months and on stable treatment regimen

Exclusion Criteria: none

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Depression symptoms | 24 weeks
  Ascertained by Beck Depression Inventory (score 0-63, higher score means worse outcome)

SECONDARY OUTCOMES:
Depression symptoms | 24 weeks
  Ascertained by Patient Health Questionnaire 9 (score 0-27, higher score means worse outcome)
Anxiety symptoms | 24 weeks
  Ascertained by Generalized Anxiety Disorder 7 (score 0-21, higher score means worse outcome)

OTHER OUTCOMES:
Negative mood deregulation | 24 weeks
  Ascertained by Negative Mood Regulation Scale (score 30-150, higher score means better outcome)
Perceived social support | 24 weeks
  Ascertained by Medical Outcomes Survey (score 0-100, higher score means better outcome)
Perceived stress | 24 weeks
  Ascertained by Perceived Stress Scale 10 (score 0-40, higher score means worse outcome)
Behavioral activation | 24 weeks
  Ascertained by Behavioral Activation for Depression Scale (score 0-150, higher score means better outcome)
Decentering | 24 weeks
  Ascertained by Experiences Questionnaire (score 20-100, higher score means better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Keshet Ronen, PhD, MPH, Principal Investigator — University of Washington
Locations (1):
- Perinatal Support Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
This project is required to deposit mental health outcomes data in the NIMH National Data Archive (NDA). NDA uses direct identifies to generate global unique identifiers, but the identifiers themselves will not be shared.
Supporting Information: SAP
Time Frame: 1/31/2027 - indefinite
Access Criteria: Data is publicly available after creating an account with the NIMH NDA
URL: https://nda.nih.gov/